CLINICAL TRIAL: NCT04279132
Title: THE EFFECT OF TOTAL INTRAVENOUS ANESTHESIA AND INHALATION ANESTHESIA TECHNIQUES FOR MINI MENTAL STATE EXAMINATION TEST AND NEURON SPECIFIC ENOLASE LEVEL IN LUMBAR DISK HERNIECTOMY OPERATIONS
Brief Title: EFFECT OF ANESTHESİA TECHNIQUES ON POSTOPERATİVE COGNİTİVE DYSFUNCTION FOR MMSE AND NSE LEVEL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, TULAY CEREN OLMEZTURK KARAKURT, MD, Erzincan University
Other Study IDs: 19/10
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Cognitive Dysfunction; NEURON SPECIFIC ENOLASE; MINI MENTAL STATE EXAMINATION TEST
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — BLOOD SAMPLES
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TOTAL INTRAVENOUS ANESTHESIA
  Interventions: Behavioral: POSTOPERATIVE COGNITIVE DYSFUNCTION
- INHALATION ANESTHESIA
  Interventions: Behavioral: POSTOPERATIVE COGNITIVE DYSFUNCTION

INTERVENTIONS:
Behavioral: POSTOPERATIVE COGNITIVE DYSFUNCTION — NEURON SPECIFIC ENOLASE LEVELS IN LUMBAR DISC HERNIECTOMY WITH GENERAL ANESTHESIA MODALITIES

SUMMARY:
The aim of this study is to compare the effects of total intravenous anesthesia and inhalation anesthesia methods on postoperative cognitive dysfunction according to Mini Mental State Examination scores and Neuron Specific Enolase levels in lumbar disc herniectomy operations.

ELIGIBILITY:
Inclusion Criteria:

-Lumbal disc herniectomy operation 18-65 age

Exclusion Criteria:

* Patients before and after the coronary artery bypass graft surgery
* patients in the last trimester of pregnancy
* patients with severe heart failure
* liver failure
* kidney failure
* malignant hyperthermia
* lactating patients
* patients with vision or hearing problems
* patients having difficulty in understanding and speaking Turkish
* Parkinson's and Alzheimer's disease
* alcohol and drug addicts
* morbidly obese patients
* intraoperative hypotension, hypertension and hypoxemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lumbal disc herniectomy operation is planned for ASA I, II and III risk group between the ages of 18-65.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-21 (Estimated); Primary Completion 2020-05-21 (Estimated); Study Completion 2020-07-21 (Estimated)

PRIMARY OUTCOMES:
MINI MENTAL STATE EXAMINATION TEST | 1 MONTH
  BELOW 27 SCORE IS ASSOSIATED WITH POSTOPERATIVE COGNITIVE DYSFUNCTION

CONTACTS AND LOCATIONS:
Overall Officials: TÜLAY CEREN ÖLMEZTÜRK KARAKURT, Principal Investigator — ERZINCAN BYU
Locations (1):
- Erzincan Byu, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goswami U, Babbar S, Tiwari S. Comparative evaluation of the effects of propofol and sevoflurane on cognitive function and memory in patients undergoing laparoscopic cholecystectomy: A randomised prospective study. Indian J Anaesth. 2015 Mar;59(3):150-5. doi: 10.4103/0019-5049.153036. PMID 25838586
- [Result] Luescher T, Mueller J, Isenschmid C, Kalt J, Rasiah R, Tondorf T, Gamp M, Becker C, Sutter R, Tisljar K, Schuetz P, Marsch S, Hunziker S. Neuron-specific enolase (NSE) improves clinical risk scores for prediction of neurological outcome and death in cardiac arrest patients: Results from a prospective trial. Resuscitation. 2019 Sep;142:50-60. doi: 10.1016/j.resuscitation.2019.07.003. Epub 2019 Jul 12. PMID 31306716
- [Result] Baysalman HB, Oğuz G, Açıkgöz G, Aksakal FN, Ünver SJJotTA, Dergisi ICS-JTAvR. Total İntravenöz ve Desfluran Anestezilerinin Erken Derlenme ve Kognitif Fonksiyonlara Etkileri. 2011;39(1).